CLINICAL TRIAL: NCT01336348
Title: Comparison of Multiple Oral and/or Intravenous Anti-platelet Strategies in Patients With ST-segment Elevation Myocardial Infarction Undergoing Primary PCI
Brief Title: Facilitation Through Aggrastat By drOpping or Shortening Infusion Line in Patients With ST-segment Elevation Myocardial Infarction Compared to or on Top of PRasugrel Loading dOse
Acronym: FABOLUS PRO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Marco Valgimigli, University of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAB-PRO-I
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: ST Segment Elevation Myocardial Infarction
Keywords: Prasugrel; Tirofiban; Clopidogrel; glycoprotein IIa/IIIa inhibitors; P2Y12 blockers
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Prasugrel Hydrochloride; Tirofiban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- prasugrel (Experimental): Prasugrel 60 mg loading dose
  Interventions: Drug: Prasugrel
- Tirofiban (Active Comparator): Tirofiban will be at a bolus only of 25uM or followed by 2 hour infusion
  Interventions: Drug: Tirofiban

INTERVENTIONS:
Drug: Prasugrel — 60 mg loading dose given orally at presentation
  Arms: prasugrel
Drug: Tirofiban — Tirofiban will be given at high bolus dose only of bolus followed by 2 H infusion in a randomized manner (1:1 ratio).
  Arms: Tirofiban

SUMMARY:
This is a single-centre, open-label prospective randomized pharmacodynamic investigation of 2 antiplatelet regimens in patients undergoing coronary intervention for ST segment elevation myocardial infarction(STEMI):

1. Tirofiban bolus only or bolus followed by 2 hour infusion on top of 600 mg clopidogrel or 60 mg prasugrel.
2. Prasugrel given at 60 mg.

DETAILED DESCRIPTION:
Primary hypothesis: Percentage IPA after 20uMol/ADP at 30' will be superior in the tirofiban arm (as aggregate) versus prasugrel alone arm Percentage IPA at 30' after 20uMol/ADP 90%±15 and 80%±15 in the tirofiban and prasugrel alone arm, respectively. For a power of 90% and an alpha error set at 5%, 50 patients per group have to be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Chest pain for >30 min with an electrocardiographic ST-segment elevation more than 1 mm in two or more contiguous electrocardiogram (ECG) leads, or with a new left bundle-branch block, and admission either within 12 h of symptom onset or between 12 and 24 h after onset with evidence of continuing ischemia

Exclusion Criteria:

* Administration of fibrinolytic or any GP IIbIIIa inhibitors for the treatment of current AMI or within 1 month before history of bleeding diathesis
* Known sensitivity to abciximab, to any component of the product or to murine monoclonal antibodies
* Major surgery or trauma within 30 days
* Active bleeding
* Previous stroke in the last six months
* Oral anticoagulant therapy
* Pre-existing thrombocytopenia
* Vasculitis
* Hypertensive retinopathy
* Severe hepatic failure
* Severe renal failure requiring haemodialysis
* Documented allergy/intolerance or contraindication to clopidogrel or inability to assume clopidogrel on a consecutive daily basis for a minimum of 30 days, or to heparin or aspirin
* Uncontrolled hypertension (systolic or diastolic arterial pressure >180 mmHg or 120, respectively, despite medical therapy)
* Limited life expectancy, e.g. neoplasms, others
* Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Percentage IPA after 20uMol/ADP at 30' will be superior in the tirofiban arm (as aggregate) versus prasugrel alone arm | 30 minutes
  Platelet aggregation (PA) will be performed as previously reported [J Am Coll Cardiol 2006;48:2178-85]. Blood samples anticoagulated with 0.129 mol/l sodium citrate will be collected for platelet reactivity. Platelet-rich plasma, obtained by centrifuging whole blood for 10 min at 200 g, will be stimulated with 5 and 20 µmol/l adenosine 5'-diphosphate (ADP) (Alfa Wasserman, Bologna, Italia) and aggregation will be assessed using a AggRAM Advanced Modular System light transmittance aggregometer.

SECONDARY OUTCOMES:
Percentage IPA at 15 minutes after ADP or TRAP induced platelet aggregation via traditional light transmission aggregometry. | 15 minutes
  Blood samples draen at 15', 30', 1H, 2H, 6H and 18-24H, anticoagulated with 0.129 mol/l sodium citrate will be collected for platelet reactivity. Platelet-rich plasma, obtained by centrifuging whole blood for 10 min at 200 g, will be stimulated with 5 and 20 µmol/l adenosine 5'-diphosphate (ADP) and 5 and 15 TRAP.
Clinical outcomes | 1 year
  Death, Myocardial infarction, stroke and the need for target vessel revascularisation will be monitored up to 1 year
Percentage IPA at 1 hour after ADP or TRAP induced platelet aggregation via traditional light transmission aggregometry. | 1 hour
  Blood samples draen at 15', 30', 1H, 2H, 6H and 18-24H, anticoagulated with 0.129 mol/l sodium citrate will be collected for platelet reactivity. Platelet-rich plasma, obtained by centrifuging whole blood for 10 min at 200 g, will be stimulated with 5 and 20 µmol/l adenosine 5'-diphosphate (ADP) and 5 and 15 TRAP.
Percentage IPA at 2 hours after ADP or TRAP induced platelet aggregation via traditional light transmission aggregometry. | 2 hours
  Blood samples draen at 15', 30', 1H, 2H, 6H and 18-24H, anticoagulated with 0.129 mol/l sodium citrate will be collected for platelet reactivity. Platelet-rich plasma, obtained by centrifuging whole blood for 10 min at 200 g, will be stimulated with 5 and 20 µmol/l adenosine 5'-diphosphate (ADP) and 5 and 15 TRAP.
Percentage IPA at 6 hours after ADP or TRAP induced platelet aggregation via traditional light transmission aggregometry. | 6 hours
  Blood samples draen at 15', 30', 1H, 2H, 6H and 18-24H, anticoagulated with 0.129 mol/l sodium citrate will be collected for platelet reactivity. Platelet-rich plasma, obtained by centrifuging whole blood for 10 min at 200 g, will be stimulated with 5 and 20 µmol/l adenosine 5'-diphosphate (ADP) and 5 and 15 TRAP.
Percentage IPA at 18-24 hours after ADP or TRAP induced platelet aggregation via traditional light transmission aggregometry. | 18-24 hours
  Blood samples draen at 15', 30', 1H, 2H, 6H and 18-24H, anticoagulated with 0.129 mol/l sodium citrate will be collected for platelet reactivity. Platelet-rich plasma, obtained by centrifuging whole blood for 10 min at 200 g, will be stimulated with 5 and 20 µmol/l adenosine 5'-diphosphate (ADP) and 5 and 15 TRAP.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Unit, Ferrara, Ferrara, Italy

REFERENCES:
- [Derived] Valgimigli M, Tebaldi M, Campo G, Gambetti S, Bristot L, Monti M, Parrinello G, Ferrari R; FABOLUS PRO Investigators. Prasugrel versus tirofiban bolus with or without short post-bolus infusion with or without concomitant prasugrel administration in patients with myocardial infarction undergoing coronary stenting: the FABOLUS PRO (Facilitation through Aggrastat By drOpping or shortening Infusion Line in patients with ST-segment elevation myocardial infarction compared to or on top of PRasugrel given at loading dOse) trial. JACC Cardiovasc Interv. 2012 Mar;5(3):268-77. doi: 10.1016/j.jcin.2012.01.006. PMID 22440491